CLINICAL TRIAL: NCT07375719
Title: Nuclear Abnormalities in Gingival Epithelial Cells in Relation to Periodontal Disease Severity and Glycemic Control
Brief Title: Nuclear Abnormalities in Gingival Epithelial Cells in Relation to Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Basak Karasu, Assist.Prof, Çankırı Karatekin University
Other Study IDs: Decision No: 11; Date: 05/02/2
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes (DM); Periodontitis; Periodontitis (Stage 3); Micronuclei Count
Keywords: diabetes; periodontitis; cytology; nuclear aberrations
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Poor Glycemic Control - Stage I-II Periodontitis: Participants with diabetes mellitus and poor glycemic control (HbA1c ≥7%) diagnosed with Stage I-II periodontitis according to the 2018 periodontal classification.
- Poor Glycemic Control - Stage III-IV Periodontitis: Participants with diabetes mellitus and poor glycemic control (HbA1c ≥7%) diagnosed with Stage III-IV periodontitis.
- Good Glycemic Control - Stage I-II Periodontitis: Participants with diabetes mellitus and good glycemic control (HbA1c <7%) diagnosed with Stage III-IV periodontitis.
- Systemically Healthy - Stage I-II Periodontitis: Systemically healthy individuals without diabetes diagnosed with Stage I-II periodontitis.
- Systemically Healthy - Stage III-IV Periodontitis: Systemically healthy individuals without diabetes diagnosed with Stage III-IV periodontitis.
- Good Glycemic Control - Stage III-IV Periodontitis: Participants with diabetes mellitus and good glycemic control (HbA1c <7%) diagnosed with Stage III-IV periodontitis.

SUMMARY:
Diabetes mellitus and periodontitis are two highly prevalent chronic diseases with a well-established bidirectional relationship. Poor glycemic control has been associated with increased periodontal inflammation and disease progression, while periodontal disease may adversely affect metabolic control in individuals with diabetes. Gingival epithelial cells, characterized by a high turnover rate, may reflect early nuclear and cellular alterations related to chronic inflammatory and metabolic conditions.

The purpose of this cross-sectional observational study is to evaluate the association between glycemic control status, determined by hemoglobin A1c (HbA1c) levels, and nuclear morphological alterations in exfoliated gingival epithelial cells in patients with diabetes mellitus presenting with different severities of periodontal disease. Nuclear biomarkers, including micronuclei formation, binucleated cells, nuclear-to-cytoplasmic (N/C) ratio alterations, and perinuclear halo formation, are assessed using cytological analysis.

Additionally, the study aims to investigate the combined and independent effects of periodontal disease severity and glycemic control on nuclear structural changes in gingival epithelial cells, comparing individuals with good (HbA1c <7%) and poor (HbA1c ≥7%) glycemic control across different periodontal stages. This study seeks to contribute to the understanding of cellular-level alterations associated with chronic periodontal inflammation and metabolic dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Diagnosis of periodontitis according to the 2018 periodontal classification
* Absence of systemic diseases other than diabetes mellitus

Exclusion Criteria:

* Presence of oral mucosal lesions
* History of malignancy
* Receipt of periodontal therapy within the previous 6 months
* Pregnancy or lactation
* Current or former tobacco use
* Alcohol consumption
* Known anemia
* Vitamin B12 deficiency
* Folate deficiency
* Presence of systemic diseases (other than diabetes mellitus) that could affect periodontal status or cellular morphology

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with DM were stratified based on glycemic control, defined by HbA1c levels, and periodontal disease severity. Accordingly, patients with poor glycemic control (HbA1c ≥7%) were classified as having Stage I-II periodontitis (Group 1, n = 14) or Stage III-IV periodontitis (Group 2, n = 18), whereas patients with good glycemic control (HbA1c <7%) were categorized as Stage I-II periodontitis (Group 3, n = 14) or Stage III-IV periodontitis (Group 4, n = 17).
  Systemically healthy individuals without diabetes served as controls and were further stratified according to periodontal disease severity, comprising Stage I-II periodontitis (Group 5, n = 16) and Stage III-IV periodontitis (Group 6, n = 16). This grouping strategy enabled assessment of both the independent and combined effects of periodontal disease severity and glycemic control on nuclear morphological alterations in gingival epithelial cells.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Nuclear morphological alterations in gingival epithelial cells | Baseline (at enrollment, single assessment)
  Quantitative assessment of nuclear morphological changes in exfoliated gingival epithelial cells, including micronuclei frequency, binucleated cells, nuclear-to-cytoplasmic (N/C) ratio alterations, and perinuclear halo formation, evaluated by light microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Üniversitesi, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical restrictions and the observational nature of the study.

REFERENCES:
- [Background] Serikova OV, Shumilovich BR, Filippova ZA, et al (2023) Nuclear aberrations in the gingival epithelium of patients with chronic periodontitis. J Indian Soc Periodontol 27:374-380. https://doi.org/10.4103/jisp.jisp_18_22
- [Background] Liu C-J, Chang W-J, Chen C-Y, et al (2015) Dynamic cellular and molecular modulations of diabetes mediated head and neck carcinogenesis. Oncotarget 6:29268-29284. https://doi.org/10.18632/oncotarget.4922
- [Background] Agrawal R, Kumar N, Gupta K, Singh TB (2018) Correlation between fasting blood sugar and cytomorphometric values of diabetic patient's buccal mucosa exfoliative cytology. J Cancer Res Ther 14:398-402. https://doi.org/10.4103/jcrt.JCRT_1211_16
- [Background] Seifi S, Feizi F, Moazzezi Z, et al (2014) Evaluation of oral mucosal epithelium in diabetic male patients by exfoliative cytology method. J Diabetes Metab Disord 13:77. https://doi.org/10.1186/2251-6581-13-77
- [Background] Bastos-Aires D, Azevedo Á, de Lurdes Pereira M, et al (2013) Preliminary study of micronuclei levels in oral exfoliated cells from patients with periodontitis. J Dent Sci 8:200-204. https://doi.org/10.1016/j.jds.2012.12.007
- [Background] Brandão P de TJ, Gomes-Filho IS, Cruz SS, et al (2015) Can periodontal infection induce genotoxic effects? Acta Odontol Scand 73:219-225. https://doi.org/10.3109/00016357.2014.982705
- [Background] Xiang D, Sun Y, Jiao C, et al (2025) Diabetes and periodontitis: the role of a high-glucose microenvironment in periodontal tissue cells and corresponding therapeutic strategies. Stem Cell Res Ther 16:366. https://doi.org/10.1186/s13287-025-04441-z
- [Background] James SL et al. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. The Lancet 392:1789-1858
- [Background] Papapanou PN, Sanz M, Buduneli N, et al (2018) Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol 89:. https://doi.org/10.1002/JPER.17
- [Background] Saravani S, Karimkoshteh A, Samaei Rahni M, Kadeh H (2021) Cytomorphometric Assessment of Buccal Mucosa Cells and Blood Sugar Status in Diabetic Patients in Zahedan (2019). Med J Islam Repub Iran. https://doi.org/10.47176/mjiri.
- [Background] Ong KL et al. (2023) Global, regional, and national burden of diabetes from 1990 to 2021, with projections of prevalence to 2050: a systematic analysis for the Global Burden of Disease Study 2021. The Lancet 402:203
- [Background] Omer MAEM, Zeen AA-AM, Ahmed HAE, et al (2025) Assessment of Micronuclei Frequency in Buccal Mucosal Cells among Diabetic Patients in Shendi, Sudan: A Cross-Sectional Case-Control Study. Saudi Journal of Medicine 10:501-506. https://doi.org/10.36348/sjm.2025.v10i10.002